CLINICAL TRIAL: NCT03418727
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter, Proof-of-Concept Study of Brimonidine Eye Drops for the Treatment of Dry Eye Disease (DED)
Brief Title: Dry Eye Disease Study With Brimonidine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCU-310-DED-2017
Record Dates: First submitted 2017-10-10; First posted 2018-02-01 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Brimonidine Tartrate; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug Arm #1 (Experimental): Combination Therapy: brimonidine (0.2%) administered as eye drops, followed by corticosteroid eye drops, two times a day (BID) for 12 weeks
  Interventions: Drug: Brimonidine; Drug: Corticosteroid Eye Drop
- Study Drug Arm #2 (Experimental): Monotherapy: brimonidine (0.2%) administered as eye drops followed by placebo, two times a day (BID) for 12 weeks
  Interventions: Drug: Brimonidine Mono Therapy
- Control Arm (Placebo Comparator): Placebo: sodium carboxymethylcellulose (0.25%) administered as eye drops followed by a second application, two time a day (BID) for 12 weeks
  Interventions: Drug: sodium carboxymethylcellulose

INTERVENTIONS:
Drug: Brimonidine — Two products delivered in sequence twice daily.
  Arms: Study Drug Arm #1
Drug: Brimonidine Mono Therapy — Brimonidine given twice daily along with placebo drops
  Arms: Study Drug Arm #2
Drug: sodium carboxymethylcellulose — Placebo given twice daily.
  Arms: Control Arm
Drug: Corticosteroid Eye Drop — Eye drop to be administered after Brimonidine in treatment arm 1
  Arms: Study Drug Arm #1

SUMMARY:
To evaluate the tolerability and preliminary efficacy of Brimonidine eye drops (with and without corticosteroid eye drops) for the treatment of Dry Eye Disease (DED).

DETAILED DESCRIPTION:
Subjects will assess their tolerance to the administration of the study drug, utilizing a Visual Analog Scale (VAS). The VAS is a 100-mm horizontal line with verbal descriptors at either end. The VAS ratings will be completed after administration of the study drug on Day 1 (post-dose), Day 28, Day 56, Day 84, and Day 105. Subjects will place a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Sign and date informed consent form approved by the IRB
3. History of Dry Eye Disease
4. Objective evidence of DED in at least one eye by having 2 or more of the following 4 signs in the same eye at Screening and Baseline (Day 1) visits:

   i. Conjunctival staining at >/= 1 (out of a possible score of 6 per eye) ii. Corneal staining at >/= 2 (out of a possible score of 15 per eye) iii. Noninvasive Tear Break-Up Time (NITBUT) at </= 7 seconds iv. Schirmer test at <10mm in 5 minutes
5. Symptomatic evidence of DED by having a global symptom score (SANDE) >/= 25 mm at both Screening and Baseline (Day 1) visits
6. Intraocular pressure (IOP) >/= 5 mmHg and </= 22 mmHg in each eye
7. Women who satisfy one of the following:

   1. Are of child-bearing potential (WOCP) who are not pregnant or lactating and who are either abstinent or sexually active on an acceptable method of birth control for at least 4 weeks prior to Visit 1 and throughout the study, OR
   2. Are post-menopausal or have undergone a sterilization procedure

Exclusion Criteria:

1. Allergic to brimonidine, corticosteroids or any similar products, or excipients of brimonidine including benzalkonium chloride (BAK)
2. Use of contact lenses
3. Currently receiving brimonidine or other treatment for glaucoma or ocular hypertension or history of glaucoma surgery.
4. Receiving or have received any experimental or investigational drug or device within 30 days prior to Screening visit
5. Intraocular pressure <5 mmHg or >22 mmHg in either eye
6. Active ocular infection or history of ocular herpetic keratitis
7. History of neurotrophic keratitis or ocular neuropathic pain
8. Any history of eyelid surgery or intraocular/ocular surgery within the past 3 months
9. Punctal occlusion within 3 months prior to Screening visit or during study
10. Corneal epithelial defect larger than 1 mm2 in either eye
11. Have active drug/alcohol dependence or abuse history
12. Are neonates, pregnant/lactating women, children, institutionalized individuals, or others who may be considered vulnerable populations
13. Received corticosteroid-containing eye drops within the past 7 days or systemic corticosteroids/immunosuppressives within the past 3 months
14. Received cyclosporine ophthalmic emulsion 0.05% (Restasis®) or lifitegrast ophthalmic solution 5% (Xiidra™) within 30 days prior to Screening visit
15. In the opinion of Investigator or Study Coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops
16. Disease, condition, or disorder that in the judgement of Investigator could confound study assessments or limit compliance to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Brenart Eye Clinic, Yorkville, Illinois
  - The Eye Institute of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Brimonidine and Corticosteroid Combination Therapy: Brimonidine (0.2%) administered as eye drops, followed by loteprednol ophthalmic suspension (0.2%), two times a day (BID) for 12 weeks
- Brimonidine Monotherapy: Brimonidine (0.2%) administered as eye drops followed by placebo BID for 12 weeks
- Placebo: Sodium carboxymethylcellulose (0.25%) administered as eye drops followed by a second application BID for 12 weeks
Period: Overall Study
Arm/Group | Brimonidine and Corticosteroid Combination Therapy | Brimonidine Monotherapy | Placebo
Started | 29 | 28 | 27
Received at Least 1 Study Treatment | 29 | 28 | 27
Completed | 28 | 26 | 25
Not Completed | 1 | 2 | 2
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized population including all participants who were randomized to the treatment
Groups:
- Brimonidine and Corticosteroid Combination Therapy: Brimonidine (0.2%) administered as eye drops, followed by loteprednol ophthalmic suspension (0.2%) BID for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Brimonidine and Corticosteroid Combination Therapy | Brimonidine Monotherapy | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 27 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.41) | 60.4 (13.88) | 59.2 (14.23) | 60.6 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 18 | 69
  Male | 3 | 3 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 5
  Not Hispanic or Latino | 29 | 25 | 25 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 28 | 27 | 26 | 81
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tolerance of Test Substance Visual Analogue Scale (VAS) Score
Description: Participants assessed their tolerance to the administration of the study drug, utilizing a VAS. The VAS is a 100-mm horizontal line with verbal descriptors at either end. Participants placed a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm).
Time Frame: Days 1, 28, 56, and 84
Population: Safety population that included all randomized participants who received at least one dose of study medication. Here, the overall number of participants analyzed are those evaluable for this Outcome Measure and the Number Analyzed per Row is the number of participants with evaluable data at each time point.
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Brimonidine and Corticosteroid Combination Therapy | Brimonidine Monotherapy | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale
  Day 1 | 82.1 [74.5 to 89.8] | 87.0 [82.2 to 91.9] | 95.0 [92.3 to 97.7]
  Day 28: number analyzed (Participants) | 28 | 28 | 24
  Day 28 | 91.1 [86.6 to 95.5] | 87.4 [82.5 to 92.3] | 88.2 [82.7 to 93.7]
  Day 56: number analyzed (Participants) | 27 | 26 | 24
  Day 56 | 92.0 [88.3 to 95.8] | 85.6 [80.6 to 90.7] | 91.0 [84.2 to 97.9]
  Day 84: number analyzed (Participants) | 28 | 25 | 25
  Day 84 | 87.8 [82.2 to 93.5] | 85.9 [78.6 to 93.1] | 94.8 [91.6 to 98.1]

ADVERSE EVENTS:
Time Frame: Day 1 (post-dose) up to 105 Days
Arm/Group | Brimonidine and Corticosteroid Combination Therapy | Brimonidine Monotherapy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/28 | 1/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine and Corticosteroid Combination Therapy (N=29) | Brimonidine Monotherapy (N=28) | Placebo (N=27)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Knee operation (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03418727/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT03418727/SAP_001.pdf